CLINICAL TRIAL: NCT00888589
Title: Improved Sensitivity for the Detection of Aggressive Breast Tumors Using 99mTc-NC100692 and a Dual-headed Small Field of View CZT Gamma Camera.
Brief Title: Detection of Aggressive Breast Tumors Using Tc-99m-NC100692
Status: Completed | Type: Observational
Sponsor: Michael O'Connor (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Michael O'Connor, Prefessor of Radiologic Physics, Mayo Clinic
Organization: Mayo Clinic (Other)
Other Study IDs: 08-001022
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer
Keywords: MBI; Molecular Breast Imaging; Breast; Breast Cancer; Molecular Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare two types of radioactive drugs to see if they provide the same or different information about any disease that may be present in the participants breast.

ELIGIBILITY:
Inclusion Criteria:

* Have a lesion on mammogram, ultrasound or breast MRI that measured < 15 mm in diameter, is considered suggestive or highly suggestive of malignancy according to the Breast Imaging Reporting and Data System Atlas criteria (BIRADS 4b, 4c or 5), and is scheduled for biopsy (needle biopsy and/or surgical biopsy).

OR

* Have a lesion on mammogram, ultrasound or breast MRI that measured > 15 mm in diameter, is known to be malignant and is scheduled for surgery.
* Patient age > 18 years of age.
* Have a negative pregnancy test on the first day of the study, or must be postmenopausal or surgically sterilized.

Exclusion Criteria:

* Patients will be excluded if they have a small lesion (< 15 mm) and have undergone prior needle biopsy of the lesion (such biopsy may effectively remove all or part of the lesion and angiogenesis associated with wound healing might confound imaging results with 99mTc-NC100692).
* Patient's pregnancy is not negative on the first day of the study, or the patient is unable to complete the pregnancy test
* Patient is unable to sit on a chair for 40 minutes

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are scheduled for a biopsy at the Mayo Clinic in Rochester, MN. The patients must have a suspicious lesion
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Evidence of disease confirmed by surgery, or benign disease confirmed by biopsy | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Judy Boughey, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] O'Connor MK, Morrow MMB, Hunt KN, Boughey JC, Wahner-Roedler DL, Conners AL, Rhodes DJ, Hruska CB. Comparison of Tc-99m maraciclatide and Tc-99m sestamibi molecular breast imaging in patients with suspected breast cancer. EJNMMI Res. 2017 Dec;7(1):5. doi: 10.1186/s13550-017-0255-6. Epub 2017 Jan 14. PMID 28091980